CLINICAL TRIAL: NCT04168450
Title: Evaluation of the Wheelchair In-Seat Activity Tracker (WiSAT)
Brief Title: Evaluation of Wheelchair In-Seat Activity Tracker
Acronym: WiSAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Georgia Institute of Technology (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patricia Karg, Associate Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: STUDY19090305; W81XWH-17-1-0221 (Other Grant/Funding Number: Department of Defense (DoD))
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Pressure Ulcer, Buttock; Pressure Injury; Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WiSAT Passive (Other): This arm is composed of participants who meet their activity threshold over the 4-week period.
  Interventions: Other: WiSAT System, Passive Feedback
- WiSAT Active (Other): This arm is composed of participants who do not meet their activity threshold over the 4-week period.
  Interventions: Other: WiSAT System, Active Feedback

INTERVENTIONS:
Other: WiSAT System, Passive Feedback — The WiSAT system is installed in the participant's wheelchair cushion and a smartphone application is installed on his/her cellphone. Participants are able to view the application as they please and they will receive no notifications from the app regarding their movement goals.
  Arms: WiSAT Passive
Other: WiSAT System, Active Feedback — The WiSAT system is installed in the participant's wheelchair cushion and smartphone application is installed on his/her cellphone. Participants receive notifications from the app to help them meet their movement goals.
  Arms: WiSAT Active

SUMMARY:
Individuals who use wheelchairs are at an increased risk of developing pressure injuries on the parts of the body that are in constant contact with the wheelchair. The development of pressure injuries can cause reduced mobility, reduced activity and participation, greater unemployment, increased risk for future pressure injury development, and premature death. There are numerous risk factors associated with developing pressure injuries. Individuals can reduce the risk of pressure injury formation by changing positions, weight-shifting, and using special cushions, but many people still struggle with pressure injuries.

This study is designed to assess the clinical effectiveness of WiSAT (Wheelchair in-Seat Activity Tracker). WiSAT is a tool designed to help prevent the development of pressure ulcers by changing behaviors that can lead to pressure ulcers. WiSAT monitors and provides real-time feedback on weight shifts and pressure relief behaviors while sitting in a wheelchair.

DETAILED DESCRIPTION:
Pressure injuries are a serious health concern for individuals who use wheelchairs. Wheelchair users are at an increased risk of developing pressure injuries on the parts of the body that are in constant contact with the wheelchair. The development of pressure injuries can cause negative consequences on their lives. Pressure injuries often lead to reduced mobility, reduced activity and participation, greater unemployment, increased risk for future pressure injury development, and premature death. Some risk factors associated with developing pressure injuries include continual pressure, nutrition, shear forces, and moisture. Individuals whose use wheelchairs can reduce the risk of pressure injury formation by changing positions, weight-shifting, and using skin protection cushions, but many people still struggle with pressure injuries.

This study will assess the clinical effectiveness and usability of WiSAT (Wheelchair in-Seat Activity Tracker). WiSAT provides real-time feedback on in-seat movement, including volitional pressure reliefs and weight-shift activity. The study's aim is to assess whether monitoring and feedback of in-seat movement can change the behavior of wheelchair users by increasing movement activities.

Study Protocol: The study will prospectively collect in-seat movement activity during everyday life for wheelchair users at risk for pressure ulcers. 25 individuals who are full-time users of wheelchairs and have a self-reported risk for pressure ulcers on the buttocks (sacrum/coccyx, ischial tuberosity, trochanter) will be recruited for the study.

Each person will have two appointments with investigators to educate, set them up with the WiSAT system and finally to remove the sensor system from the cushion.

The first visit will take approximately 1.5 to 2 hours, in which participants will provide written informed consent. During this visit, demographic and clinical information will be collected via self-report. All participants will then receive education about skin health including information about pressure ulcers, prevention strategies such as pressure relieving techniques in both bed and wheelchair, and the importance of checking skin regularly for signs of pressure issues. The WiSAT hardware will be placed within the cover and beneath their current wheelchair cushion to measure and transmit baseline seat movement activity; with no mobile application and visual feedback initiated at this time. Subjects' baseline behavior will be monitored for two weeks to serve as the comparator for the enabled WiSAT system.

After 14 days of baseline monitoring, the app will automatically switch to feedback mode. Participants will be informed that they can now monitor their movement activity. Each subject will be given the ability to set his or her own goals using the app settings. The movement activity feedback will be provided passively for four weeks, requiring them to view the application on their smartphone to see daily movement activity data.

After the four weeks of app use, recorded movement activity will be used to categorize participants as meeting or not meeting the movement threshold. Subjects who do not attain their movement threshold will be provided with active feedback using audible and/or haptic reminders. Those who have reached their threshold will continue to access the app to review their activity (passive feedback).

All participants will be followed for a total of 2.5 months: 2 weeks baseline, 4 weeks passive visual feedback only, and 4 weeks of passive and/or active feedback. At the end of the study, the team will collect feedback on usability and acceptability of the activity tracker.

ELIGIBILITY:
Inclusion Criteria:

* Use a wheelchair as their primary means of mobility
* Have a self-reported history of pressure ulcers on the buttocks within the past three years
* Age 18 or older
* Use a smartphone with an operating system upgraded in the last 5 years
* Use a skin protection cushion or skin protection/positioning cushion

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average daily movement activity at 5 months | baseline (2 weeks) and 5 months
  Average daily movement activity is defined as the frequency of in-seat movement will be calculated as total number of weight shifts and pressure reliefs per unit time of wheelchair use (movements/hour).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia E Karg, MS, Study Director — University of Pittsburgh
Locations (2):
- United States (2):
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified research data may in the future be shared upon request with investigators external to the study team who are conducting similar research with an approved IRB. Research data including time in wheelchair, weight shift frequency, and demographics may be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Any time after primary and secondary publications
Access Criteria: To be determined.